CLINICAL TRIAL: NCT03682757
Title: Post-Injury Platelet Biology: Mechanisms and Outcomes
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Colorado, Denver (Other); University of Utah (Other); University of California, Berkeley (Other); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: P0528296; 5K23GM130892 (NIH)
Record Dates: First submitted 2018-09-17; First posted 2018-09-25 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Wound and Injuries; Blood Platelets; Endothelium
Keywords: Trauma; Platelets; Coagulopathy
MeSH Terms: conditions — Wounds and Injuries; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Severe Injury/Shock: Severely injured trauma patients presenting with shock, as defined by an Injury Severity Score (ISS)>=25, and base deficit (BD)>=6.
- Without Severe Injury/Shock: Not severely injured trauma patients presenting without shock, as defined by an Injury Severity Score (ISS)<25, and base deficit (BD) <6.
- Healthy Controls: Uninjured healthy volunteers

SUMMARY:
Trauma-induced coagulopathy is a central cause of preventable deaths from hemorrhage after injury. The contribution and impact of altered post injury platelet biology on trauma-induced coagulopathy is not well understood despite the pivotal contribution of platelets to normal coagulation and endothelial integrity. The central hypothesis for this study is that severe injury and shock drive altered platelet activation, platelet aggregation, and platelet-endothelial interactions that are associated with increased rates of transfusion, organ failure, and mortality. This study will investigate these causal pathways, mechanisms, and associated outcomes in a prospective observational trauma cohort through collection of biospecimens and detailed clinical data.

DETAILED DESCRIPTION:
This is a prospective cohort study of trauma patients on admission to the emergency department and for the subsequent 28 days. All adult patients meeting criteria for full trauma team activation and admitted to Zuckerberg San Francisco General Hospital and Trauma center, a level-1 trauma center, are eligible for enrollment. A 20-ml sample of blood will be drawn within 10 minutes of arrival in the emergency department (ED), processed in the central laboratory, and plasma stored at -80°C. Blood samples will be collected immediately on presentation via initial placement of a 16-gauge or larger peripheral intravenous line. Plasma biomarkers of endothelial injury will be measured by enzyme-linked immunosorbent assays (von Willebrand factor, syndecan-1, and angiopoietin-2). Cellular biomarkers of platelet activation will be measured by flow cytometry (platelet-monocyte aggregates, integrin αIIbβ3, P-selectin, and platelet microparticles). Platelet aggregation will be measured by whole blood multiple electrode impedance aggregometry. The effect of post-injury platelets on endothelial integrity will be quantified by in vitro assays of platelet-induced endothelial permeability. Comprehensive demographic data and medical history will be collected from chart review, interviews of patients and family members. Detailed clinical and outcome data is collected including transfusion timing and doses, the incidence of organ failure (Denver Postinjury Multiple Organ Failure Score), acute respiratory distress syndrome (Berlin Definition), infection, symptomatic thromboembolic complications, ventilator-free days, length of intensive care unit (ICU) and hospital stay, and mortality (6 hours, 24 hours, 30 days). In hospital mortality after 30 days will be assessed for all patients. Standard coagulation measures (international normalized ratio, prothrombin time, platelet count) and other laboratory measures will be collected to account and control for other distinct but highly integrated pathways implicated in trauma-induced coagulopathy. The Trauma Registry, a large database managed under guidelines from the American Trauma society, uses chart review to retrospectively assign Injury Severity Scores (ISS) and Abbreviated Injury Scores (AIS).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients meeting criteria for full trauma team activation and admitted to Zuckerberg San Francisco General Hospital.

Exclusion Criteria:

* Patients <18 years old
* Patients transferred from other hospitals
* Patients who are pregnant
* Patients who are incarcerated
* Patients will be retrospectively excluded if they were taking anticoagulant or anti-platelet medications, have moderate or severe liver disease, or a known bleeding diathesis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients meeting criteria for full trauma team activation and admitted to Zuckerberg San Francisco General Hospital
Sampling Method: Non-Probability Sample
Enrollment: 367 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
In Vitro Measurement of Endothelial Biomarkers | 0 hour (within 10 minutes of arrival to the Emergency Department)
  Plasma biomarkers of endothelial injury will be measured by enzyme-linked immunosorbent assays (von Willebrand factor, syndecan-1, and angiopoietin-2).
In Vitro Measurement Platelet Activation Biomarkers | 0 hour (within 10 minutes of arrival to the Emergency Department)
  Cellular biomarkers of platelet activation will be measured by flow cytometry (platelet-monocyte aggregates, integrin αIIbβ3, P-selectin, and platelet microparticles).
In Vitro Measurement of Platelet Aggregation | 0 hour (within 10 minutes of arrival to the Emergency Department)
  Platelet aggregation will be measured by whole blood multiple electrode impedance aggregometry.
In Vitro Assays of Platelet-Induced Endothelial Permeability | 0 hour (within 10 minutes of arrival to the Emergency Department)
  The effect of post-injury platelets on endothelial integrity will be quantified by in vitro assays of platelet-induced endothelial permeability using transendothelial permeability electrical resistance (TEER) assays.
Transfusion products received (red cell, plasma, platelet) | in first 24 hours after arrival to the emergency department
  Continuous units of red cell, plasma, platelet; transfused in 24 hours (yes/no); massive transfusion (>10units red cell/24 hour, yes/no)
Organ Failure | Within 1 week of arrival to the emergency department
  Rates of organ failure (yes/no) (Denver Postinjury Multiple Organ Failure Score)
6-hour Mortality | 6 hours after arrival to the emergency department
24-hour Mortality | 24 hours after arrival to the emergency department
30-days Mortality | 30 days after arrival to the emergency department
Hospital Discharge Mortality | Through hospital discharge (an average of 13 days)

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Kornblith, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Norton R, Kobusingye O. Injuries. N Engl J Med. 2013 May 2;368(18):1723-30. doi: 10.1056/NEJMra1109343. No abstract available. PMID 23635052
- [Background] Cannon JW. Hemorrhagic Shock. N Engl J Med. 2018 Jan 25;378(4):370-379. doi: 10.1056/NEJMra1705649. No abstract available. PMID 29365303
- [Background] Kauvar DS, Lefering R, Wade CE. Impact of hemorrhage on trauma outcome: an overview of epidemiology, clinical presentations, and therapeutic considerations. J Trauma. 2006 Jun;60(6 Suppl):S3-11. doi: 10.1097/01.ta.0000199961.02677.19. PMID 16763478
- [Background] Cohen MJ, Christie SA. New understandings of post injury coagulation and resuscitation. Int J Surg. 2016 Sep;33(Pt B):242-245. doi: 10.1016/j.ijsu.2016.05.037. Epub 2016 May 19. PMID 27212591
- [Background] Brohi K, Singh J, Heron M, Coats T. Acute traumatic coagulopathy. J Trauma. 2003 Jun;54(6):1127-30. doi: 10.1097/01.TA.0000069184.82147.06. PMID 12813333
- [Background] MacLeod JB, Lynn M, McKenney MG, Cohn SM, Murtha M. Early coagulopathy predicts mortality in trauma. J Trauma. 2003 Jul;55(1):39-44. doi: 10.1097/01.TA.0000075338.21177.EF. PMID 12855879
- [Background] Baimukanova G, Miyazawa B, Potter DR, Gibb SL, Keating S, Danesh A, Beyer A, Dayter Y, Bruhn R, Muench MO, Cap AP, Norris PJ, Spinella P, Cohen M, Pati S. The effects of 22 degrees C and 4 degrees C storage of platelets on vascular endothelial integrity and function. Transfusion. 2016 Mar;56 Suppl 1:S52-64. doi: 10.1111/trf.13455. PMID 27001362
- [Background] Baimukanova G, Miyazawa B, Potter DR, Muench MO, Bruhn R, Gibb SL, Spinella PC, Cap AP, Cohen MJ, Pati S. Platelets regulate vascular endothelial stability: assessing the storage lesion and donor variability of apheresis platelets. Transfusion. 2016 Mar;56 Suppl 1(Suppl 1):S65-75. doi: 10.1111/trf.13532. PMID 27001364
- [Background] Kutcher ME, Redick BJ, McCreery RC, Crane IM, Greenberg MD, Cachola LM, Nelson MF, Cohen MJ. Characterization of platelet dysfunction after trauma. J Trauma Acute Care Surg. 2012 Jul;73(1):13-9. doi: 10.1097/TA.0b013e318256deab. PMID 22743367
- [Background] Davenport RA, Brohi K. Coagulopathy in trauma patients: importance of thrombocyte function? Curr Opin Anaesthesiol. 2009 Apr;22(2):261-6. doi: 10.1097/ACO.0b013e328325a6d9. PMID 19390252
- [Background] Brown LM, Call MS, Margaret Knudson M, Cohen MJ; Trauma Outcomes Group; Holcomb JB, Wade CE, Brasel KJ, Vercruysse G, MacLeod J, Dutton RP, Hess JR, Duchesne JC, McSwain NE, Muskat P, Johannigamn J, Cryer HM, Tillou A, Pittet JF, De Moya MA, Schreiber MA, Tieu B, Brundage S, Napolitano LM, Brunsvold M, Brunsvold M, Beilman G, Peitzman AB, Zenait MS, Sperry J, Alarcon L, Croce MA, Minei JP, Kozar R, Gonzalez EA, Stewart RM, Cohn SM, Mickalek JE, Bulger EM, Cotton BA, Nunez TC, Ivatury R, Meredith JW, Miller P, Pomper GJ, Marin B. A normal platelet count may not be enough: the impact of admission platelet count on mortality and transfusion in severely injured trauma patients. J Trauma. 2011 Aug;71(2 Suppl 3):S337-42. doi: 10.1097/TA.0b013e318227f67c. PMID 21814101
- [Background] Kornblith LZ, Kutcher ME, Redick BJ, Calfee CS, Vilardi RF, Cohen MJ. Fibrinogen and platelet contributions to clot formation: implications for trauma resuscitation and thromboprophylaxis. J Trauma Acute Care Surg. 2014 Feb;76(2):255-6; discussion 262-3. doi: 10.1097/TA.0000000000000108. PMID 24458031
- [Background] Li R, Elmongy H, Sims C, Diamond SL. Ex vivo recapitulation of trauma-induced coagulopathy and preliminary assessment of trauma patient platelet function under flow using microfluidic technology. J Trauma Acute Care Surg. 2016 Mar;80(3):440-9. doi: 10.1097/TA.0000000000000915. PMID 27082706
- [Background] Wohlauer MV, Moore EE, Thomas S, Sauaia A, Evans E, Harr J, Silliman CC, Ploplis V, Castellino FJ, Walsh M. Early platelet dysfunction: an unrecognized role in the acute coagulopathy of trauma. J Am Coll Surg. 2012 May;214(5):739-46. doi: 10.1016/j.jamcollsurg.2012.01.050. PMID 22520693
- [Background] Jacoby RC, Owings JT, Holmes J, Battistella FD, Gosselin RC, Paglieroni TG. Platelet activation and function after trauma. J Trauma. 2001 Oct;51(4):639-47. doi: 10.1097/00005373-200110000-00003. PMID 11586152
- [Background] Briggs A, Gates JD, Kaufman RM, Calahan C, Gormley WB, Havens JM. Platelet dysfunction and platelet transfusion in traumatic brain injury. J Surg Res. 2015 Feb;193(2):802-6. doi: 10.1016/j.jss.2014.08.016. Epub 2014 Aug 13. PMID 25218281
- [Background] Nachman RL, Rafii S. Platelets, petechiae, and preservation of the vascular wall. N Engl J Med. 2008 Sep 18;359(12):1261-70. doi: 10.1056/NEJMra0800887. No abstract available. PMID 18799560
- [Background] Fiedler U, Scharpfenecker M, Koidl S, Hegen A, Grunow V, Schmidt JM, Kriz W, Thurston G, Augustin HG. The Tie-2 ligand angiopoietin-2 is stored in and rapidly released upon stimulation from endothelial cell Weibel-Palade bodies. Blood. 2004 Jun 1;103(11):4150-6. doi: 10.1182/blood-2003-10-3685. Epub 2004 Feb 19. PMID 14976056
- [Background] Kozar RA, Pati S. Syndecan-1 restitution by plasma after hemorrhagic shock. J Trauma Acute Care Surg. 2015 Jun;78(6 Suppl 1):S83-6. doi: 10.1097/TA.0000000000000631. No abstract available. PMID 26002270
- [Background] Peng Z, Pati S, Potter D, Brown R, Holcomb JB, Grill R, Wataha K, Park PW, Xue H, Kozar RA. Fresh frozen plasma lessens pulmonary endothelial inflammation and hyperpermeability after hemorrhagic shock and is associated with loss of syndecan 1. Shock. 2013 Sep;40(3):195-202. doi: 10.1097/SHK.0b013e31829f91fc. PMID 23807246
- [Background] Naumann DN, Hazeldine J, Davies DJ, Bishop J, Midwinter MJ, Belli A, Harrison P, Lord JM. Endotheliopathy of Trauma is an on-Scene Phenomenon, and is Associated with Multiple Organ Dysfunction Syndrome: A Prospective Observational Study. Shock. 2018 Apr;49(4):420-428. doi: 10.1097/SHK.0000000000000999. PMID 28945676
- [Background] Rodriguez EG, Ostrowski SR, Cardenas JC, Baer LA, Tomasek JS, Henriksen HH, Stensballe J, Cotton BA, Holcomb JB, Johansson PI, Wade CE. Syndecan-1: A Quantitative Marker for the Endotheliopathy of Trauma. J Am Coll Surg. 2017 Sep;225(3):419-427. doi: 10.1016/j.jamcollsurg.2017.05.012. Epub 2017 Jun 1. PMID 28579548
- [Background] Zipperle J, Altenburger K, Ponschab M, Schlimp CJ, Spittler A, Bahrami S, Redl H, Schochl H. Potential role of platelet-leukocyte aggregation in trauma-induced coagulopathy: Ex vivo findings. J Trauma Acute Care Surg. 2017 May;82(5):921-926. doi: 10.1097/TA.0000000000001410. PMID 28257393
- [Background] Michelson AD, Barnard MR, Hechtman HB, MacGregor H, Connolly RJ, Loscalzo J, Valeri CR. In vivo tracking of platelets: circulating degranulated platelets rapidly lose surface P-selectin but continue to circulate and function. Proc Natl Acad Sci U S A. 1996 Oct 15;93(21):11877-82. doi: 10.1073/pnas.93.21.11877. PMID 8876231
- [Background] Michelson AD, Barnard MR, Krueger LA, Valeri CR, Furman MI. Circulating monocyte-platelet aggregates are a more sensitive marker of in vivo platelet activation than platelet surface P-selectin: studies in baboons, human coronary intervention, and human acute myocardial infarction. Circulation. 2001 Sep 25;104(13):1533-7. doi: 10.1161/hc3801.095588. PMID 11571248
- [Background] Rondina MT, Grissom CK, Men S, Harris ES, Schwertz H, Zimmerman GA, Weyrich AS. Whole blood flow cytometry measurements of in vivo platelet activation in critically-Ill patients are influenced by variability in blood sampling techniques. Thromb Res. 2012 Jun;129(6):729-35. doi: 10.1016/j.thromres.2011.11.031. Epub 2011 Dec 16. PMID 22178064
- [Background] Murray CJ, Lopez AD. Mortality by cause for eight regions of the world: Global Burden of Disease Study. Lancet. 1997 May 3;349(9061):1269-76. doi: 10.1016/S0140-6736(96)07493-4. PMID 9142060
- [Background] Scope A, Farkash U, Lynn M, Abargel A, Eldad A. Mortality epidemiology in low-intensity warfare: Israel Defense Forces' experience. Injury. 2001 Jan;32(1):1-3. doi: 10.1016/s0020-1383(00)00101-7. PMID 11164393
- [Background] Baker SP, Whitfield RA, O'Neill B. Geographic variations in mortality from motor vehicle crashes. N Engl J Med. 1987 May 28;316(22):1384-7. doi: 10.1056/NEJM198705283162206. PMID 3574414
- [Background] Hess JR, Brohi K, Dutton RP, Hauser CJ, Holcomb JB, Kluger Y, Mackway-Jones K, Parr MJ, Rizoli SB, Yukioka T, Hoyt DB, Bouillon B. The coagulopathy of trauma: a review of mechanisms. J Trauma. 2008 Oct;65(4):748-54. doi: 10.1097/TA.0b013e3181877a9c. PMID 18849786
- [Background] White NJ, Ward KR, Pati S, Strandenes G, Cap AP. Hemorrhagic blood failure: Oxygen debt, coagulopathy, and endothelial damage. J Trauma Acute Care Surg. 2017 Jun;82(6S Suppl 1):S41-S49. doi: 10.1097/TA.0000000000001436. PMID 28328671
- [Background] Stansbury LG, Hess AS, Thompson K, Kramer B, Scalea TM, Hess JR. The clinical significance of platelet counts in the first 24 hours after severe injury. Transfusion. 2013 Apr;53(4):783-9. doi: 10.1111/j.1537-2995.2012.03828.x. Epub 2012 Aug 6. PMID 22882316
- [Background] Davis PK, Musunuru H, Walsh M, Cassady R, Yount R, Losiniecki A, Moore EE, Wohlauer MV, Howard J, Ploplis VA, Castellino FJ, Thomas SG. Platelet dysfunction is an early marker for traumatic brain injury-induced coagulopathy. Neurocrit Care. 2013 Apr;18(2):201-8. doi: 10.1007/s12028-012-9745-6. PMID 22847397
- [Background] Donahue DL, Beck J, Fritz B, Davis P, Sandoval-Cooper MJ, Thomas SG, Yount RA, Walsh M, Ploplis VA, Castellino FJ. Early platelet dysfunction in a rodent model of blunt traumatic brain injury reflects the acute traumatic coagulopathy found in humans. J Neurotrauma. 2014 Feb 15;31(4):404-10. doi: 10.1089/neu.2013.3089. Epub 2013 Nov 21. PMID 24040968
- [Background] Bhandari V, Choo-Wing R, Lee CG, Zhu Z, Nedrelow JH, Chupp GL, Zhang X, Matthay MA, Ware LB, Homer RJ, Lee PJ, Geick A, de Fougerolles AR, Elias JA. Hyperoxia causes angiopoietin 2-mediated acute lung injury and necrotic cell death. Nat Med. 2006 Nov;12(11):1286-93. doi: 10.1038/nm1494. Epub 2006 Nov 5. PMID 17086189
- [Background] Calfee CS, Gallagher D, Abbott J, Thompson BT, Matthay MA; NHLBI ARDS Network. Plasma angiopoietin-2 in clinical acute lung injury: prognostic and pathogenetic significance. Crit Care Med. 2012 Jun;40(6):1731-7. doi: 10.1097/CCM.0b013e3182451c87. PMID 22610178
- [Background] Ong T, McClintock DE, Kallet RH, Ware LB, Matthay MA, Liu KD. Ratio of angiopoietin-2 to angiopoietin-1 as a predictor of mortality in acute lung injury patients. Crit Care Med. 2010 Sep;38(9):1845-51. doi: 10.1097/CCM.0b013e3181eaa5bf. PMID 20581666
- [Background] Pati S, Potter DR, Baimukanova G, Farrel DH, Holcomb JB, Schreiber MA. Modulating the endotheliopathy of trauma: Factor concentrate versus fresh frozen plasma. J Trauma Acute Care Surg. 2016 Apr;80(4):576-84; discussion 584-5. doi: 10.1097/TA.0000000000000961. PMID 26808040
- [Background] Potter DR, Baimukanova G, Keating SM, Deng X, Chu JA, Gibb SL, Peng Z, Muench MO, Fomin ME, Spinella PC, Kozar R, Pati S. Fresh frozen plasma and spray-dried plasma mitigate pulmonary vascular permeability and inflammation in hemorrhagic shock. J Trauma Acute Care Surg. 2015 Jun;78(6 Suppl 1):S7-S17. doi: 10.1097/TA.0000000000000630. PMID 26002267
- [Background] Naumann DN, Hazeldine J, Dinsdale RJ, Bishop JR, Midwinter MJ, Harrison P, Hutchings SD, Lord JM. Endotheliopathy is associated with higher levels of cell-free DNA following major trauma: A prospective observational study. PLoS One. 2017 Dec 19;12(12):e0189870. doi: 10.1371/journal.pone.0189870. eCollection 2017. PMID 29261771
- [Background] Johansson PI, Henriksen HH, Stensballe J, Gybel-Brask M, Cardenas JC, Baer LA, Cotton BA, Holcomb JB, Wade CE, Ostrowski SR. Traumatic Endotheliopathy: A Prospective Observational Study of 424 Severely Injured Patients. Ann Surg. 2017 Mar;265(3):597-603. doi: 10.1097/SLA.0000000000001751. PMID 27144442
- [Background] Brohi K, Cohen MJ, Ganter MT, Matthay MA, Mackersie RC, Pittet JF. Acute traumatic coagulopathy: initiated by hypoperfusion: modulated through the protein C pathway? Ann Surg. 2007 May;245(5):812-8. doi: 10.1097/01.sla.0000256862.79374.31. PMID 17457176
- [Background] Moore FA, Sauaia A, Moore EE, Haenel JB, Burch JM, Lezotte DC. Postinjury multiple organ failure: a bimodal phenomenon. J Trauma. 1996 Apr;40(4):501-10; discussion 510-2. doi: 10.1097/00005373-199604000-00001. PMID 8614027
- [Background] Sauaia A, Moore FA, Moore EE, Lezotte DC. Early risk factors for postinjury multiple organ failure. World J Surg. 1996 May;20(4):392-400. doi: 10.1007/s002689900062. PMID 8662125
- [Background] Sauaia A, Moore EE, Johnson JL, Ciesla DJ, Biffl WL, Banerjee A. Validation of postinjury multiple organ failure scores. Shock. 2009 May;31(5):438-47. doi: 10.1097/SHK.0b013e31818ba4c6. PMID 18838942
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Rondina MT, Carlisle M, Fraughton T, Brown SM, Miller RR 3rd, Harris ES, Weyrich AS, Zimmerman GA, Supiano MA, Grissom CK. Platelet-monocyte aggregate formation and mortality risk in older patients with severe sepsis and septic shock. J Gerontol A Biol Sci Med Sci. 2015 Feb;70(2):225-31. doi: 10.1093/gerona/glu082. Epub 2014 Jun 10. PMID 24917177
- [Background] Shih L, Kaplan D, Kraiss LW, Casper TC, Pendleton RC, Peters CL, Supiano MA, Zimmerman GA, Weyrich AS, Rondina MT. Platelet-Monocyte Aggregates and C-Reactive Protein are Associated with VTE in Older Surgical Patients. Sci Rep. 2016 Jun 7;6:27478. doi: 10.1038/srep27478. PMID 27270163
- [Background] Solomon C, Traintinger S, Ziegler B, Hanke A, Rahe-Meyer N, Voelckel W, Schochl H. Platelet function following trauma. A multiple electrode aggregometry study. Thromb Haemost. 2011 Aug;106(2):322-30. doi: 10.1160/TH11-03-0175. Epub 2011 Jun 9. PMID 21655681
- [Background] Ding N, Chen G, Hoffman R, Loughran PA, Sodhi CP, Hackam DJ, Billiar TR, Neal MD. Toll-like receptor 4 regulates platelet function and contributes to coagulation abnormality and organ injury in hemorrhagic shock and resuscitation. Circ Cardiovasc Genet. 2014 Oct;7(5):615-24. doi: 10.1161/CIRCGENETICS.113.000398. Epub 2014 Jul 21. PMID 25049041
- [Background] Sapru A, Calfee CS, Liu KD, Kangelaris K, Hansen H, Pawlikowska L, Ware LB, Alkhouli MF, Abbott J, Matthay MA; NHLBI ARDS Network. Plasma soluble thrombomodulin levels are associated with mortality in the acute respiratory distress syndrome. Intensive Care Med. 2015 Mar;41(3):470-8. doi: 10.1007/s00134-015-3648-x. Epub 2015 Feb 3. PMID 25643902
- [Background] Ware LB, Fang X, Matthay MA. Protein C and thrombomodulin in human acute lung injury. Am J Physiol Lung Cell Mol Physiol. 2003 Sep;285(3):L514-21. doi: 10.1152/ajplung.00442.2002. Epub 2003 May 16. PMID 12754194
- [Background] Weyrich AS, Denis MM, Kuhlmann-Eyre JR, Spencer ED, Dixon DA, Marathe GK, McIntyre TM, Zimmerman GA, Prescott SM. Dipyridamole selectively inhibits inflammatory gene expression in platelet-monocyte aggregates. Circulation. 2005 Feb 8;111(5):633-42. doi: 10.1161/01.CIR.0000154607.90506.45. Epub 2005 Jan 24. PMID 15668340